CLINICAL TRIAL: NCT05770687
Title: Real World Observation of SGLT2 Inhibitors on Clinical Outcomes and Left Ventricular Remodeling in Type 2 Diabetic Patients with Acute Myocardial Infarction, a Prospective, Multi-center Registry Study
Brief Title: SGLT2 Inhibitors on Clinical Outcomes and Left Ventricular Remodeling in Type 2 Diabetic Patients with Acute Myocardial Infarction, a Prospective, Multi-center Registry Study
Acronym: RECORD-AMI
Status: Recruiting | Type: Observational
Sponsor: Kiyuk Chang (Other)
Collaborators: Seoul St. Mary's Hospital (Other); Uijeongbu St. Mary Hospital (Other); Incheon St.Mary's Hospital (Other); Daejeon St. Mary's hospital (Other); Bucheon St. Mary's Hospital (Other); St Vincent's Hospital (Other); Yeouido St. Mary's Hospital (Other); Sejong General Hospital (Other); Pusan National University Hospital (Other); Andong Hospital (Unknown); Chungnam National University Hospital (Other); St. Carollo General Hospital (Unknown); Pusan National University Yangsan Hospital (Other); Kyungpook National University Hospital (Other); Jeju National University Hospital (Other); Korea University Anam Hospital (Other); Inje University (Other)
Responsible Party: Sponsor-Investigator, Kiyuk Chang, MD, PhD, Seoul St. Mary's Hospital
Organization: Seoul St. Mary's Hospital (Other)
Other Study IDs: KC19OEDI0591
Record Dates: First submitted 2023-03-05; First posted 2023-03-15 (Actual); Last update posted 2025-01-03 (Actual); Status verified 2025-01

CONDITIONS: Myocardial Infarction; Diabetes Mellitus, Type 2
Keywords: Percutaneous Coronary Intervention; SGLT-2 inhibitor
MeSH Terms: conditions — Myocardial Infarction; Diabetes Mellitus, Type 2 | interventions — Sodium-Glucose Transporter 2 Inhibitors; dapagliflozin; empagliflozin; ertugliflozin; ipragliflozin

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- SGLT-2 inhibitor: Patients with naive use of SGLT-2 inhibitors after PCI
  Interventions: Drug: SGLT2 inhibitor

INTERVENTIONS:
Drug: SGLT2 inhibitor — Patients started on SGLT2 inhibitors after PCI for AMI
  Other Names: dapagliflozin, empagliflozin, ertugliflozin, ipragliflozin

SUMMARY:
Prospective trials performed on type 2 diabetes patients without established cardiovascular disease has shown that SGLT2 inhibitors reduce cardiovascular risk. No studies have yet examined the occurrence of cardiovascular disease in patients with acute myocardial infarction.

The investigators designed the current study to evaluate the most ideal oral hypoglycemic agent in type 2 diabetes patients undergoing percutaneous coronary intervention for acute myocardial infarction. The investigators hypothesize that the use of SGLT-2 inhibitors will reduce cardiovascular events and modify left ventricular remodeling after myocardial infarctions.

DETAILED DESCRIPTION:
8 hospitals of the Catholic University of Korea with high-volume percutaneous coronary intervention of following hospitals are participating in the current study.

Seoul St. Mary's Hospital, Seoul, South Korea

Yeoido St. Mary's Hospital, Seoul, South Korea

Uijongbu St. Mary's Hospital, Gyeonggi-do, South Korea

Eunpyeong St. Mary's Hospital, Seoul, South Korea

Bucheon St. Mary's Hospital, Gyeonggi-do, South Korea

Incheon St. Mary's Hospital, Incheon, South Korea

St. Vincent Hospital, Gyeonggi-do, South Korea

Daejeon St. Mary's Hospital, Daejeon, South Korea

After recruitment of all patients, the control group will be selected from a previous prospective cohort (COREA-AMI, NCT02385682) using identical inclusion / exclusion criteria except for use of SGLT2 inhibitors. The control cohort of 3,000 patients will be selected using 1:3 propensity matching.

ELIGIBILITY:
Inclusion Criteria:

* Acute myocardial infarction who were treated with percutaneous coronary intervention
* Type 2 diabetes mellitus
* Started SGLT2 inhibitors <1 month before/after PCI

Exclusion Criteria:

* Type 1 diabetes mellitus
* Insulin / GLP-1 analogue users
* Previous users of SGLT2 inhibitors
* Pregnancy

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Type 2 diabetes mellitus patients undergoing percutaneous coronary intervention for acute myocardial infarction
Sampling Method: Non-Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2020-08-01 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Major adverse cardiac and cerebrovascular events | 2 years
  A composite of cardiac death, nonfatal MI, nonfatal stroke, and HF hospitalization

SECONDARY OUTCOMES:
Cardiac death | 2 years
  Cardiovascular death
Nonfatal myocardial infarction | 2 years
  non-fatal myocardial infarction
Nonfatal stroke | 2 years
  non-fatal stroke
Hospitalization for heart failure | 2 years
  hospitalization for HF
Target lesion revascularization | 2 years
  Revascularization performed for target lesion
Target vessel revascularization | 2 years
  Revascularization performed for target vessel
Non-target vessel revascularization | 2 years
  Revascularization performed for non-target vessel
Definite/Probable stent thrombosis | 2 years
  Definite or probable stent thrombosis
Absolute and percentage change of microalbuminuria | 2 years
  Absolute and percentage change of microalbuminuria
Absolute and percentage change of HbA1c | 2 years
  Absolute and percentage change of HbA1c
Absolute and percentage change of NT-proBNP | 2 years
  Absolute and percentage change of NT-proBNP
Absolute and percentage change of BMI | 2 years
  Absolute and percentage change of BMI
Absolute and percentage change of body weight | 2 years
  Absolute and percentage change of body weight
Changes in echocardiograhic parameters | 1 year
  LVEF, LVEDV, LVESV, LVMI, E, A, DT, E/E'

CONTACTS AND LOCATIONS:
Overall Officials: Kiyuk Chang, MD, PhD, Principal Investigator — Seoul St. Mary's Hospital
Locations (1):
- Seoul St. Mary's Hospital, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No